CLINICAL TRIAL: NCT02167750
Title: Effects of Phytochemicals on Aspects of Cognitive Performance
Brief Title: Effect of Phytochemicals on Aspects of Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1404
Record Dates: First submitted 2014-06-10; First posted 2014-06-19 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Performance
Keywords: cognitive; phytochmicals; caffeine; cognitive performance after ingestion of test beverage

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cherry flavored beverage - Mix 1 (Placebo Comparator): Mix 1 flavored still beverage
  Interventions: Other: Cherry Flavored Beverage
- Cherry Flavored Beverage - Mix 2 (Experimental): Mix 2 flavored still beverage with phytochmicals and caffeine
  Interventions: Other: Cherry Flavored Beverage
- Cherry Flavored Beverage - Mix 3 (Experimental): Mix 3 flavored still beverage with phytochemicals and caffeine
  Interventions: Other: Cherry Flavored Beverage
- Cherry Flavored Beverage - Mix 4 (Experimental): Mix 4 flavored still beverage with phytochemicals and caffeine
  Interventions: Other: Cherry Flavored Beverage
- Cherry Flavored Beverage - Mix 5 (Experimental): Mix 5 flavored still beverage with phytochemicals and caffeine
  Interventions: Other: Cherry Flavored Beverage
- Cherry Flavored Beverage - Mix 6 (Experimental): Mix 6 flavored still beverage with caffeine
  Interventions: Other: Cherry Flavored Beverage

INTERVENTIONS:
Other: Cherry Flavored Beverage — Intervention involves consuming one beverage at the beginning of each visit of the crossover sequence.

SUMMARY:
The primary purpose of the research is to test the short-term effects of the consumption of beverages containing phytochemicals and caffeine on several aspects of cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be older than 17 and under 50 years of age, self report of good health

Exclusion Criteria:

* Using any prescription medication including birth control;
* Report a history of any phschiatric condition;
* Report hypersinsitivity to caffeine;
* Have visual impairment that connot be corrected with glasses or contact lenses

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the changes in the ratings from computer administered tasks within the domains of mood, short-term recognition memory, and attention from pre- to post-study product consumption and between treatment conditions | 0-80 minutes post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Univerysity of Georgia, Athens, Georgia, United States